CLINICAL TRIAL: NCT04183556
Title: The Effect of Turmeric on New Onset Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batman Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erhan Okuyan,M.D, Obstetrician and gynaecologist, Batman Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BatmanMCHH
Record Dates: First submitted 2019-11-24; First posted 2019-12-03 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Primary Dysmenorrhea
Keywords: new onset primary dysmenorrhea; turmeric; naproxen
MeSH Terms: interventions — Naproxen; Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1/NSAI(nonsteroidal anti-inflammatory agent) group (Active Comparator): Patients with naproxen drug therapy for early onset dysmenorrhea.
  Interventions: Drug: Naproxen
- 2/NSAI+ Turmeric (1 gram oral powder formula per day ) (Placebo Comparator): NSAI(nonsteroidal anti-inflammatory agent) + Turmeric for early onset dysmenorrhea (1 gram oral powder formula in mens time)
  Interventions: Drug: Naproxen; Dietary Supplement: Turmeric

INTERVENTIONS:
Drug: Naproxen — use of naproxen twice a day orally in mens time
  Other Names: NSAI(nonsteroidal anti-inflammatory agent)
Dietary Supplement: Turmeric — Use of turmeric orally (1 gram powder formula) in mens time
  Arms: 2/NSAI+ Turmeric (1 gram oral powder formula per day )

SUMMARY:
The study was planned as 150 patients. Patients who met early-onset dysmenorrhea criteria and who met the inclusion criteria; 150 patients were divided into 2 equal groups, and NSAID during the menstrual cycle, nsai + turmeric 1 gr oral powder form treatment was planned to be started in the other group. The pain frequency and severity before and after treatment were evaluated by visual analog scale and the two groups were compared.

DETAILED DESCRIPTION:
There are scientific publications on the use of turmeric, which constitutes the hypothesis of our study, in branches such as cardiology, neurology, infertility and chest diseases due to its anti-inflammatory, anti-aging properties.

The data are planned to be evaluated by the researchers using the SPSS(Statistical Package for the Social Sciences ) 17.0 program on computer. The responses of all groups to the VAS scores are planned to be entered into the system by using the SPSS program before and after treatment. statistics (number, percentage, mean, standard deviation), chi-square and logistic regression analysis are used to compare categorical variables. Chi-square test and Mann Whitney-U test are planned to be used in comparison between groups.When examining the difference between the groups, if the p value is less than 0.05, it is planned as a proof of significant difference.

ELIGIBILITY:
Inclusion Criteria:

1. Early-onset primary dysmenorrhea (Definition: Pain that begins in less than 6 months, is not accompanied by infection, begins on the first day of menstruation and ends on the last day of menstruation)
2. Non-pregnant and breastfeeding patients
3. Between 16-35 years old
4. No anatomic pathology or disease
5. Lack of active infection
6. No history of drug use
7. BMI is less than 25
8. Those who wish to participate in the study signed the consent form
9. Smoking, non-alcoholic patients
10. Patients who completed their treatment and came to the control
11. Regular menstruation

Exclusion Criteria:

1. Presence of vaginal infection such as Trichomonas vaginalis and candida albicans
2. Patients who do not want to participate in the study
3. Pregnant and nursing patients
4. Be under 16 years or older than 30 years
5. Systemic disease
6. Smoking, alcohol consumption
7. BMI higher than 25
8. People with organic pelvic pathology (ovarian cyst, fibroids, polyps)
9. People with a history of drug use
10. Patients who discontinue treatment and do not come to control
11. Irregular menstruation
12. Any history of contraindication to naproxen
13. Turmeric allergy history

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
the effect of turmeric on visual analog scala at new onset primary dysmenorrhea | 6 months
  To determine the effect of turmeric use on pain severity in early onset primary .The minimum pain score for dysmenorrhea is defined as 1 maximal pain score of 10 and a significant difference is planned if there is a significant difference between pretreatment scores and post-treatment scores if at least 50 percent reduction in turmeric use is achieved.It is predicted that there is no significant difference in visual analog scale scoring less than 50 percent and treatment is not effective.
  Before and after the treatment of turmeric effect on visual analog scores will be compared and a significant difference will be observed if at least 50 percent improvement is detected.dysmenorrhea using visual analogue scoring.
  The percentage of reduction in visual analog scores will be calculated in all patients using turmeric.

CONTACTS AND LOCATIONS:
Overall Officials: erhan okuyan, Principal Investigator — Batman Training and Research Hospital
Locations (1):
- Batman Maternity and Child's health Hospital, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No